CLINICAL TRIAL: NCT04161456
Title: Preliminary Efficacy and Safety of Apremilast in the Treatment of Acne Conglobata: A Phase II, Single Centre, Open Label, Proof of Concept Study for the Treatment of Acne Conglobata With the PDE-4 Inhibitor Apremilast (APACCO-Study)
Brief Title: Preliminary Efficacy and Safety of Apremilast in the Treatment of Acne Conglobata
Acronym: APACCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Frank Behrens (Other)
Collaborators: Dermatology Department University Hospital Frankfurt (Unknown); Celgene (Industry)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, Sponsor representative, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMP-0517
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Acne Conglobata
Keywords: Acne conglobata; Phosphodiesterase (PDE)-Inhibitor
MeSH Terms: conditions — Acne Conglobata | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Patients will be treated with Apremilast
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apremilast (Experimental): Apremilast twice daily 30 mg
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast twice daily 30 mg
  Other Names: Otezla

SUMMARY:
Apremilast mediates its clinical effect through the cAMP-PKA-NFkappaB pathway which results in a clinical picture changes to a decrease of all signs of inflammation.

Due to the NFkappaB mediated chronical inflammation in the pathogenesis of acne conglobata, a treatment with Apremilast seems to be an effective option.

In this study, treatment with Apremilast (Otezla®) will be performed in patients with acne conglobata to observe its preliminary efficacy and safety in an open label, single-centre proof of concept study design.

DETAILED DESCRIPTION:
Treatment options for acne conglobata are limited and those which are effective can only be used in short term such as systemic steroids, antibiotics or retinoids due to their association to side effects or potentially teratogenetic effects.

Apremilast, a specific inhibitor for PDE-4, mediates its clinical effect through the cAMP-PKA-NFkappaB pathway which results in a decrease of pro-inflammatory and increase of anti-inflammatory cytokines in several types of leukocytes. The clinical picture changes to a decrease of all signs of inflammation.

Due to the NFkappaB mediated chronical inflammation in the pathogenesis of acne conglobata, a treatment with Apremilast seems to be an effective option.

In this study, treatment with Apremilast (Otezla®) will be performed in patients with acne conglobata to observe its preliminary efficacy and safety in an open label, single-centre proof of concept study design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acne conglobata for a minimum of 6 months
* Active condition of acne conglobata, defined as minimum IGA of 2 (5-point scale) of severity of acne conglobate
* No clinical significant or severe abnormality of skin (e.g. scars, other severe skin disease) based on medical/medication history or physical examination as determined by the treating physician
* Number of abscesses ≤ 2
* Written informed consent obtained from the patients prior to the initiation of any protocol-required procedures
* Compliance to study procedures and study protocol
* Age 18 - 65 years
* patients who do not tolerate or no longer tolerate therapies or for whom the following treatment options are contraindicated:

  * Topical retinoid therapy
  * isotretinoin and/or acitretin as standard therapy
  * Topical treatment with antibiotics, glucocorticoids, retinoids, Vit-D-analogue, calcineurin inhibitors
  * systemic antibiotics, systemic glucocorticoids
  * systemic retinoids

Exclusion Criteria:

* Previous use of Apremilast, or any other PDE-4 inhibitor
* According to Summary of Product characteristics (SmPC); see special warnings regarding suicidal ideation and behaviour
* Known hypersensitivity to any component of the investigator medicinal product (IMP)
* Current use of strong CYP3A4 enzyme inducers (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin, and St. John's Wort) Active dermatologic conditions which may confound the diagnosis of acne conglobata or would interfere with the assessment of treatment (e.g., acne inversa, atopic dermatitis, seborrheic dermatitis, ichthyosis, and psoriasis)
* History of clinically significant infection within the last 4 weeks before screening, which, in the opinion of the treating physician, may compromise the safety of the patient
* Presentation of special type of acne, including but not limited to:

  * Medication related acne (e.g., steroid abuse)
  * Acne with facial edema
  * Recalcitrant acne
  * Acne cosmetic, pomade acne
  * Acne mechanica
  * Chloracne
* History of any kind of cancer or carcinoma in situ within the last 5 years before screening
* History of chronic alcohol/drug abuse within the last 12 months before screening
* Pregnant or breastfeeding women
* Females of childbearing potential not willing to use effective contraception (defined as PEARL index <1 - e.g. hormonal contraceptive containing estrogen and progesterone, or progesterone only, applied orally, intravaginal, transdermal or to be injected, IUD) for the duration of the study including also strict abstinence, or partner had a vasectomy
* Severe kidney insufficiency (glomerular filtration rate (GFR) < 30 ml/min)
* Any severe disease, which, in the opinion of the treating physician, may interfere or worsen the acne conglobata or could become a safety problem for patients
* History of or current Hepatitis-B, Hepatitis-C or HIV infection
* Any active medication which suppresses the immune system, including disease modifying anti-rheumatic drugs (DMARDs) and biologicals
* Current participation in another investigational clinical trial or participation within 30 days prior to screening
* Major surgery within the last 4 weeks before screening
* Subject susceptible to take a local corticosteroid treatment (class I - III) during the study except inhaled or topic when needed to treat a condition outside the treatment area (head, neck, upper trunk)
* History and current status of suicidal thoughts or behaviour or previous suicidal attempt
* Washout times for previous therapy for acne conglobata before screening:

  * 1 week for any topical treatment (e.g., antibiotics, glucocorticoids, retinoids, Vit-D-analogue, calcineurin inhibitors)
  * 4 weeks for any systemic antibiotics, systemic glucocorticoids or UV-therapy
  * 12 weeks for any systemic retinoids or any investigational drug
  * Patients who take any kind of contraceptive therapy (eg. estrogen, gestagen) with known positive effect on acne must be on stable dosage for a minimum of 6 month
* Underage or incapable patients
* Patients who are legally institutionalized

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
50% reduction in number of lesion | 24 weeks
  proportion of subjects who achieve at least a 50% reduction in total number of inflammatory lesions

SECONDARY OUTCOMES:
Proportionof subjects in Investigator global assessment (IGA) | Baseline to visit 3 (week 2)
  proportion of subjects who achieve an IGA 0 / 1 or an improvement of a minimum 2 points on an IGA 5-point scale (value 0 to 4, whereby 0 is symptom-free and 4 severe symptoms)
proportion of subjects in Investigator global assessment (IGA) | Baseline to visit 4 (week 4)
  proportion of subjects who achieve an IGA 0 / 1 or an improvement of a minimum 2 points on an IGA 5-point scale (value 0 to 4, whereby 0 is symptom-free and 4 severe symptoms)
proportion of subjects in Investigator global assessment (IGA) | Baseline to visit 5 (week 8)
  proportion of subjects who achieve an IGA 0 / 1 or an improvement of a minimum 2 points on an IGA 5-point scale (value 0 to 4, whereby 0 is symptom-free and 4 severe symptoms)
proportion of subjects in Investigator global assessment (IGA) | Baseline to visit 6 (week 16)
  proportion of subjects who achieve an IGA 0 / 1 or an improvement of a minimum 2 points on an IGA 5-point scale (value 0 to 4, whereby 0 is symptom-free and 4 severe symptoms)
proportion of subjects in Investigator global assessment (IGA) | Baseline to visit 7 (week 24)
  proportion of subjects who achieve an IGA 0 / 1 or an improvement of a minimum 2 points on an IGA 5-point scale (value 0 to 4, whereby 0 is symptom-free and 4 severe symptoms)
change in skin condition | at visit 3 (week 2)
  skin condition measured in Symptoms Score REduction Index (SSRI), calculated as the percentage of lesions after treatment in relation to before treatment. The lower the value the more reduction of lesions was achieved by treatment
change in skin condition | at visit 4 (week 4)
  skin condition measured in Symptoms Score REduction Index (SSRI)calculated as the percentage of lesions after treatment in relation to before treatment. The lower the value the more reduction of lesions was achieved by treatment
change in skin condition | at visit 5 (week 8)
  skin condition measured in Symptoms Score Reduction Index (SSRI)calculated as the percentage of lesions after treatment in relation to before treatment. The lower the value the more reduction of lesions was achieved by treatment
change in skin condition | at visit 6 (week 16)
  skin condition measured in Symptoms Score Reduction Index (SSRI)calculated as the percentage of lesions after treatment in relation to before treatment. The lower the value the more reduction of lesions was achieved by treatment
change in skin condition | at visit 7 (week 24)
  skin condition measured in Symptoms Score Reduction Index (SSRI)calculated as the percentage of lesions after treatment in relation to before treatment. The lower the value the more reduction of lesions was achieved by treatment
change in pain of the inflammatory lesions | at visit 3 (week 2)
  pain of the inflammatory lesions measured by a visual analog scale (VAS), measured in mm values (0 mm to 100 mm). The higher the value the more pain is experienced by the subject.
change in pain of the inflammatory lesions | at visit 4 (week 4)
  pain of the inflammatory lesions measured by a visual analog scale (VAS)measured in mm values (0 mm to 100 mm). The higher the value the more pain is experienced by the subject.
change in pain of the inflammatory lesions | at visit 5 (week 8)
  pain of the inflammatory lesions measured by a visual analog scale (VAS)measured in mm values (0 mm to 100 mm). The higher the value the more pain is experienced by the subject.
change in pain of the inflammatory lesions | at visit 6 (week 16)
  pain of the inflammatory lesions measured by a visual analog scale (VAS)measured in mm values (0 mm to 100 mm). The higher the value the more pain is experienced by the subject.
change in pain of the inflammatory lesions | at visit 7 (week 24)
  pain of the inflammatory lesions measured by a visual analog scale (VAS)measured in mm values (0 mm to 100 mm). The higher the value the more pain is experienced by the subject.
change in itch of the inflammatory lesions measured by a VAS | at visit 3 (week 2)
  itch of the inflammatory lesions measured by a VAS, measured in mm values (0 mm to 100 mm). The higher the value the more itching is experienced by the subject.
change in itch of the inflammatory lesions measured by a VAS | at visit 4 (week 4)
  itch of the inflammatory lesions measured by a VAS, measured in mm values (0 mm to 100 mm). The higher the value the more itching is experienced by the subject.
change in itch of the inflammatory lesions measured by a VAS | at visit 5 (week 8)
  itch of the inflammatory lesions measured by a VAS, measured in mm values (0 mm to 100 mm). The higher the value the more itching is experienced by the subject.
change in itch of the inflammatory lesions measured by a VAS | at visit 6 (week 16)
  itch of the inflammatory lesions measured by a VAS, measured in mm values (0 mm to 100 mm). The higher the value the more itching is experienced by the subject.
change in itch of the inflammatory lesions measured by a VAS | at visit 7 (week 24)
  itch of the inflammatory lesions measured by a VAS, measured in mm values (0 mm to 100 mm). The higher the value the more itching is experienced by the subject.
change in quality of life | Baseline to visit 3 (week 2)
  change in quality of life measured by Dermatology Life Quality Index (DLQI). The DLQI is calculated by summing the score of each of the 10 questions resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
change in quality of life | Baseline to visit 4 (week 4)
  change in quality of life measured by Dermatology Life Quality Index (DLQI).The DLQI is calculated by summing the score of each of the 10 questions resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
change in quality of life | Baseline to visit 5 (week 8)
  change in quality of life measured by Dermatology Life Quality Index (DLQI). The DLQI is calculated by summing the score of each of the 10 questions resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
change in quality of life | Baseline to visit 6 (week 16)
  change in quality of life measured by Dermatology Life Quality Index (DLQI). The DLQI is calculated by summing the score of each of the 10 questions resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
change in quality of life | Baseline to visit 7 (week 24)
  change in quality of life measured by Dermatology Life Quality Index (DLQI). The DLQI is calculated by summing the score of each of the 10 questions resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
change in depression profile | Baseline to Visit 3 (week 2)
  change in depression profile measured by Patient Health Questionnaire (PHQ-9). The PHQ-9 is the 9-item depression module from the full PHQ. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9-items can be scored from 0 (not at all) to 3 (nearly every day).
change in depression profile | Baseline to Visit 4 (week 4)
  change in depression profile measured by Patient Health Questionnaire (PHQ-9). The PHQ-9 is the 9-item depression module from the full PHQ. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9-items can be scored from 0 (not at all) to 3 (nearly every day).
change in depression profile | Baseline to Visit 5 (week 8)
  change in depression profile measured by Patient Health Questionnaire (PHQ-9).The PHQ-9 is the 9-item depression module from the full PHQ. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9-items can be scored from 0 (not at all) to 3 (nearly every day).
change in depression profile | Baseline to Visit 6 (week 16)
  change in depression profile measured by Patient Health Questionnaire (PHQ-9). The PHQ-9 is the 9-item depression module from the full PHQ. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9-items can be scored from 0 (not at all) to 3 (nearly every day).
change in depression profile | Baseline to Visit 7 (week 24)
  change in depression profile measured by Patient Health Questionnaire (PHQ-9). The PHQ-9 is the 9-item depression module from the full PHQ. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9-items can be scored from 0 (not at all) to 3 (nearly every day).
compliance to therapy (drug accountability) | at visit 3 (week 2)
  compliance to therapy measured by drug accountability (counting of returned IMP)
compliance to therapy (drug accountability) | at visit 4 (week 4)
  compliance to therapy measured by drug accountability (counting of returned IMP)
compliance to therapy (drug accountability) | at visit 5 (week 8)
  compliance to therapy measured by drug accountability (counting of returned IMP)
compliance to therapy (drug accountability) | at visit 6 (week 16)
  compliance to therapy measured by drug accountability (counting of returned IMP)
compliance to therapy (drug accountability) | at visit 7 (week 24)
  compliance to therapy measured by drug accountability (counting of returned IMP)
Frequency of adverse events (AEs) | at visit 3 (week 2)
  Frequency of adverse events (AEs) as documented in Case Report Form (CRF)
Frequency of adverse events (AEs) | at visit 4 (week 4)
  Frequency of adverse events (AEs) as documented in Case Report Form (CRF)
Frequency of adverse events (AEs) | at visit 5 (week 8)
  Frequency of adverse events (AEs) as documented in Case Report Form (CRF)
Frequency of adverse events (AEs) | at visit 6 (week 16)
  Frequency of adverse events (AEs) as documented in Case Report Form (CRF)
Frequency of adverse events (AEs) | at visit 7 (week 24)
  Frequency of adverse events (AEs) as documented in Case Report Form (CRF)
Frequency of adverse events (AEs) | at Follow-up (week 28)
  Frequency of adverse events (AEs) as documented in Case Report Form (CRF)
Seriousness of adverse events (AEs) | at visit 3 (week 2)
  Determination of seriousness of adverse events (AEs) and rate of seriousness as documented in Case Report Form (CRF)
Seriousness of adverse events (AEs) | at visit 4 (week 4)
  Determination of seriousness of adverse events (AEs) and rate of seriousness as documented in Case Report Form (CRF)
Seriousness of adverse events (AEs) | at visit 5 (week 8)
  Determination of seriousness of adverse events (AEs) and rate of seriousness as documented in Case Report Form (CRF)
Seriousness of adverse events (AEs) | at visit 6 (week 18)
  Determination of seriousness of adverse events (AEs) and rate of seriousness as documented in Case Report Form (CRF)
Seriousness of adverse events (AEs) | at visit 7 (week 24)
  Determination of seriousness of adverse events (AEs) and rate of seriousness as documented in Case Report Form (CRF)
Seriousness of adverse events (AEs) | at Follow-up (week 28)
  Determination of seriousness of adverse events (AEs) and rate of seriousness as documented in Case Report Form (CRF)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pinter, MD, Principal Investigator — University Hospital of Goethe-University Frankfurt
Locations (1):
- University Hospital Frankfurt, Frankfurt, Hessia, Germany

IPD SHARING:
Plan to Share IPD: No